CLINICAL TRIAL: NCT00954590
Title: CONTACT: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Six-Month Safety and Efficacy Study of Dimebon in Patients With Moderate-to-Severe Alzheimer's Disease
Brief Title: A Safety and Efficacy Study Evaluating Dimebon (Latrepirdine) in Patients With Moderate to Severe Alzheimer's Disease
Acronym: CONTACT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIM19
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Moderate to Severe Alzheimer
MeSH Terms: interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dimebon (latrepirdine) (Experimental): Dimebon, 20 mg orally three times daily
  Interventions: Drug: Dimebon (latrepirdine)
- Placebo (Placebo Comparator): Placebo orally three times daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimebon (latrepirdine) — 20 mg orally three times daily
  Arms: Dimebon (latrepirdine)
Drug: Placebo — Placebo orally three times daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Dimebon is safe and effective in patients with moderate to severe Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-Severe Alzheimer's disease
* Mini-Mental State Examination (MMSE) Score between 5 to 14, inclusive
* Stable on donepezil for at least 6 months

Exclusion Criteria:

* Other causes of dementia
* Major structural brain disease
* Unstable medical condition or significant hepatic or renal disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | 26 weeks post baseline
  To evaluate the efficacy of dimebon (latrepirdine) as compared to placebo on a measure of behavior, the Neuropsychiatric Inventory (NPI)
Activities of Daily Living (severe) (ADCS ADLsev) | 26 weeks post baseline
  To evaluate the efficacy of dimebon as compared to placebo on a measure of self-care and daily function, the Alzheimer's Disease Cooperative Study - Activities of Daily Living (severe) (ADCS ADLsev).

CONTACTS AND LOCATIONS:
Locations (2):
- Santiago, Chile
- Glasgow, Scotland, United Kingdom